CLINICAL TRIAL: NCT03369847
Title: Initiating Inhaled Corticosteroid Therapy at Discharge From the Pediatric Emergency Department to Prevent Asthma Relapse: A Randomized Control Trial
Brief Title: Inhaled Steroids for Pediatric Asthma at Pediatric Emergency Medicine Discharge
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-10-161-202(HHC)
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Asthma; Pediatric ALL
Keywords: inhaled corticosteroids; budesonide; beclomethasone
MeSH Terms: conditions — Asthma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Budesonide; Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Corticosteroids (Experimental): * Patients under 5 years of age will receive low dose budesonide solution 0.25mg/respule to be given twice a day via nebulizer x 28 days.
  * Patients 5 years and older will receive one beclomethasone metered-dose inhaler (MDI) 40mcg/puff two puffs twice a day via spacer x 28 days
  Interventions: Drug: budesonide, beclomethasone
- Standard Care (No Intervention): Patients allocated to this group will not receive an asthma controller medication from the emergency department. The intervention group will receive prescriptions for inhaled albuterol and oral corticosteroids as per standard treatment.

INTERVENTIONS:
Drug: budesonide, beclomethasone — The inhaled corticosteroids we are using for this study are budesonide nebulized solution and beclomethasone metered-dose inhaler. Low-doses for these medications are 0.5mg/day for budesonide and 160 mcg/day for beclomethasone. Patients under 5 years of age will receive low dose budesonide solution 0.25mg/respule to be given twice a day via nebulizer. Budesonide is FDA approved for children under 5 years of age. Patients 5 years and older will receive one beclomethasone metered-dose inhaler (MDI) 40mcg/puff two puffs twice a day via spacer. Beclomethasone is FDA approved for children 5 years and older.
  Other Names: Pulmicort, QVAR
  Arms: Inhaled Corticosteroids

SUMMARY:
This study evaluates the initiation of inhaled corticosteroids upon discharge from the pediatric emergency room in children under 18 presenting with asthma exacerbation. Half of the patients will receive a prescription for inhaled corticosteroids in addition to standard care, and half of the patients will receive standard card alone.

DETAILED DESCRIPTION:
The primary objective is to determine the effect of prescribing inhaled corticosteroids in addition to short acting beta agonists and oral corticosteroids (if indicated) from the Pediatric Emergency Department (PED) on relapse rates within 28 days. Secondary objectives include the effect of this intervention on hospitalization rates and asthma quality of life within the study period.

Selection criteria include patients aged ≤18 years presenting with a chief complaint consistent with asthma exacerbation with previous diagnosis of asthma by a physician OR one major in the Asthma Predictive Index (API) with two prior episodes of wheezing in the past year. Children who received oral corticosteroids as part of treatment during this visit for acute asthma exacerbation and deemed well enough after interventions to be discharged by the treating physician will be approached for enrollment. Exclusion criteria include patients who received asthma controller medications within four weeks prior to presentation or an allergy to intervention asthma controller mediations.

Patients will be randomized using a random number generator to the intervention group, or standard care (control) group in a 1:1 ratio. Patients assigned to the intervention group will be subject to initiation of an asthma controller medication upon discharge. The intervention group will receive a one-month supply of a low-dose inhaled corticosteroid from the PED. Patients <5 years of age or patients who prefer nebulized medications will receive a one month supply of low dose Pulmicort (budesonide) solution 0.25mg/respule to be given twice a day via nebulizer. Patients ≥5 years of age will receive one low dose QVAR (Beclometasone dipropionate) metered-dose inhaler (MDI) 40mcg/puff with instructions to take it two puffs twice a day with spacer. Patients allocated to the control group will not receive an asthma controller medication from the PED. Both groups will receive prescriptions for oral corticosteroids as per standard treatment and inhaled albuterol. The Mini Pediatric Asthma Control Tool (MPACT), a validated questionnaire used to rapidly identify persistent asthma symptoms in the PED will also be administered prior to discharge to assess for persistent asthma symptoms.

Patients will be followed up with a telephone call at 28 days to collect outcome data. Additional attempts will be made at 29 and 30 days post-discharge if initial attempts at contact are unsuccessful. Primary and secondary outcomes will be assessed during this call. The caller will not be blinded to group assignment. Asthma relapse rates, hospital admission rates, and medication compliance will be assessed during this follow up call. In addition, the Mini Pediatric Asthma Control Tool will be re-administered to assess change in asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint consistent with asthma exacerbation
* Previous diagnosis of asthma by a physician OR one major in the Asthma Predictive Index (API) with two prior episodes of wheezing in the past year.
* Major criteria in the API: parent with asthma, patient with eczema, evidence of sensitization to allergens in the air
* Received oral corticosteroids as part of treatment during this visit for acute asthma exacerbation.
* Deemed well enough after interventions to be discharged by the treating physician.
* If <5 years of age, possession of nebulizer machine at home.

Exclusion Criteria:

* Received asthma controller medications within four weeks prior to presentation
* Allergy to intervention asthma controller medications.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbation relapse | 28 days after index emergency department visit
  Emergency department/urgent care visit or unscheduled primary care doctor visit for asthma symptoms

SECONDARY OUTCOMES:
Hospital admission | 28 days after index emergency department visit
  Hospital admission
Change in Asthma control | 28 days after index emergency department visit
  Intermittent vs. persistent symptoms after the study period via repeat of the Mini Pediatric Asthma Control Tool (MPACT) score
Medication compliance | 28 days after index emergency department visit
  If prescribed an inhaled corticosteroid, defined as correct use of asthma controller medications on 80% of days

CONTACTS AND LOCATIONS:
Locations (1):
- Kings County Hospital Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] McCarren M, McDermott MF, Zalenski RJ, Jovanovic B, Marder D, Murphy DG, Kampe LM, Misiewicz VM, Rydman RJ. Prediction of relapse within eight weeks after an acute asthma exacerbation in adults. J Clin Epidemiol. 1998 Feb;51(2):107-18. doi: 10.1016/s0895-4356(97)00246-1. PMID 9474071
- [Background] Cloutier MM, Hall CB, Wakefield DB, Bailit H. Use of asthma guidelines by primary care providers to reduce hospitalizations and emergency department visits in poor, minority, urban children. J Pediatr. 2005 May;146(5):591-7. doi: 10.1016/j.jpeds.2004.12.017. PMID 15870660
- [Background] Navaratnam P, Jayawant SS, Pedersen CA, Balkrishnan R. Physician adherence to the national asthma prescribing guidelines: evidence from national outpatient survey data in the United States. Ann Allergy Asthma Immunol. 2008 Mar;100(3):216-21. doi: 10.1016/S1081-1206(10)60445-0. PMID 18426140
- [Background] Singh AK, Woodruff PG, Ritz RH, Mitchell D, Camargo CA Jr. Inhaled corticosteroids for asthma: are ED visits a missed opportunity for prevention? Am J Emerg Med. 1999 Mar;17(2):144-7. doi: 10.1016/s0735-6757(99)90047-5. PMID 10102313
- [Background] Zorc JJ, Chew A, Allen JL, Shaw K. Beliefs and barriers to follow-up after an emergency department asthma visit: a randomized trial. Pediatrics. 2009 Oct;124(4):1135-42. doi: 10.1542/peds.2008-3352. Epub 2009 Sep 28. PMID 19786448
- [Background] Andrews AL, Teufel RJ 2nd, Basco WT Jr. Initiating inhaled steroid treatment for children with asthma in the emergency room: current reported prescribing rates and frequently cited barriers. Pediatr Emerg Care. 2013 Sep;29(9):957-62. doi: 10.1097/PEC.0b013e3182a219d0. PMID 23974712
- [Background] Cydulka RK, Tamayo-Sarver JH, Wolf C, Herrick E, Gress S. Inadequate follow-up controller medications among patients with asthma who visit the emergency department. Ann Emerg Med. 2005 Oct;46(4):316-22. doi: 10.1016/j.annemergmed.2004.12.024. PMID 16187464
- [Background] Garro AC, Asnis L, Merchant RC, McQuaid EL. Frequency of prescription of inhaled corticosteroids to children with asthma in U.S. emergency departments. Acad Emerg Med. 2011 Jul;18(7):767-70. doi: 10.1111/j.1553-2712.2011.01117.x. PMID 21762239
- [Background] Scarfone RJ, Zorc JJ, Angsuco CJ. Emergency physicians' prescribing of asthma controller medications. Pediatrics. 2006 Mar;117(3):821-7. doi: 10.1542/peds.2005-0962. PMID 16510663
- [Background] Rowe BH, Bota GW, Fabris L, Therrien SA, Milner RA, Jacono J. Inhaled budesonide in addition to oral corticosteroids to prevent asthma relapse following discharge from the emergency department: a randomized controlled trial. JAMA. 1999 Jun 9;281(22):2119-26. doi: 10.1001/jama.281.22.2119. PMID 10367823
- [Background] Sin DD, Man SF. Low-dose inhaled corticosteroid therapy and risk of emergency department visits for asthma. Arch Intern Med. 2002 Jul 22;162(14):1591-5. doi: 10.1001/archinte.162.14.1591. PMID 12123402
- [Background] Sung L, Osmond MH, Klassen TP. Randomized, controlled trial of inhaled budesonide as an adjunct to oral prednisone in acute asthma. Acad Emerg Med. 1998 Mar;5(3):209-13. doi: 10.1111/j.1553-2712.1998.tb02614.x. PMID 9523927
- [Background] Andrews AL, Teufel RJ 2nd, Basco WT Jr, Simpson KN. A cost-effectiveness analysis of inhaled corticosteroid delivery for children with asthma in the emergency department. J Pediatr. 2012 Nov;161(5):903-7. doi: 10.1016/j.jpeds.2012.05.015. Epub 2012 Jun 18. PMID 22717219
- [Background] Lehman HK, Lillis KA, Shaha SH, Augustine M, Ballow M. Initiation of maintenance antiinflammatory medication in asthmatic children in a pediatric emergency department. Pediatrics. 2006 Dec;118(6):2394-401. doi: 10.1542/peds.2006-0871. PMID 17142524
- [Background] Brenner BE, Chavda KK, Camargo CA Jr. Randomized trial of inhaled flunisolide versus placebo among asthmatic patients discharged from the emergency department. Ann Emerg Med. 2000 Nov;36(5):417-26. doi: 10.1067/mem.2000.110824. PMID 11054193
- [Background] Edmonds ML, Milan SJ, Brenner BE, Camargo CA Jr, Rowe BH. Inhaled steroids for acute asthma following emergency department discharge. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD002316. doi: 10.1002/14651858.CD002316.pub2. PMID 23235590
- [Background] Topal E, Gucenmez OA, Harmanci K, Arga M, Derinoz O, Turktas I. Potential predictors of relapse after treatment of asthma exacerbations in children. Ann Allergy Asthma Immunol. 2014 Apr;112(4):361-4. doi: 10.1016/j.anai.2014.01.025. Epub 2014 Feb 28. PMID 24583137
- [Background] Castro-Rodriguez JA, Holberg CJ, Wright AL, Martinez FD. A clinical index to define risk of asthma in young children with recurrent wheezing. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1403-6. doi: 10.1164/ajrccm.162.4.9912111. PMID 11029352
- [Background] Sampayo EM, Chew A, Zorc JJ. Make an M-PACT on asthma: rapid identification of persistent asthma symptoms in a pediatric emergency department. Pediatr Emerg Care. 2010 Jan;26(1):1-5. doi: 10.1097/PEC.0b013e3181c32e9d. PMID 20042916
- [Background] Gorelick MH, Stevens MW, Schultz TR, Scribano PV. Performance of a novel clinical score, the Pediatric Asthma Severity Score (PASS), in the evaluation of acute asthma. Acad Emerg Med. 2004 Jan;11(1):10-8. doi: 10.1197/j.aem.2003.07.015. PMID 14709423
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372